CLINICAL TRIAL: NCT01222494
Title: Measurement of Cardiometabolic Risk in Antipsychotic-Treated Children
Brief Title: Healthy Bodies, Healthy Kids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-0425; K23MH092435 (NIH)
Record Dates: First submitted 2010-10-05; First posted 2010-10-18 (Estimated); Results first posted 2018-10-15 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Child Mental Disorders; Obesity; Metabolic Syndrome
Keywords: Child Psychiatry; Obesity; Antipsychotic
MeSH Terms: conditions — Neurodevelopmental Disorders; Obesity; Metabolic Syndrome | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Antipsychotic Treated Educational Cntrl (Placebo Comparator): Antipsychotic treated participants randomized to this arm will receive diet and exercise education at monthly intervals with a study clinician or coordinator.
  Interventions: Behavioral: Diet and Exercise Education
- Antipsychotic Treated Weekly BWL (Experimental): Antipsychotic treated participants randomized to this arm will engage in an evidence-based, 16 week manualized behavioral weight loss intervention that includes weekly meetings and phone check-ins with a trained study therapist.
  Interventions: Behavioral: Behavioral Weight Loss
- Non-antipsychotic Treated Weekly BWL (Active Comparator): Participants assigned to this arm will engage in an evidence-based, 16 week manualized behavioral weight loss intervention that includes weekly meetings and phone check-ins with a trained study therapist.
  Interventions: Behavioral: Behavioral Weight Loss

INTERVENTIONS:
Behavioral: Behavioral Weight Loss — This intervention is a family-based, behavioral weight loss program that has been employed in studies with overweight and obese children, as well as with children who have diabetes. For the proposed study, the program has been modified to fit the needs of disruptive and behaviorally disturbed youth and their families. The modified program includes 16 weeks of weekly visits with a study interventionist, and supplemental phone contacts as needed. Phone contacts will only replace in-person visits if absolutely necessary to achieve the visit.
  Arms: Antipsychotic Treated Weekly BWL; Non-antipsychotic Treated Weekly BWL
Behavioral: Diet and Exercise Education — Participants assigned to this arm will receive monthly medically validated, individualized diet and exercise education by a trained research professional.
  Arms: Antipsychotic Treated Educational Cntrl

SUMMARY:
The US prevalence of childhood-onset obesity and type 2 diabetes, both predictors of cardiovascular risk, have increased to epidemic proportions in recent decades. Children with mental illness, especially those treated with antipsychotic medications, are at additional risk for obesity (adiposity) and related risk conditions. A variety of noninvasive techniques to assess cardiometabolic risk have begun to be applied in children, including body composition measured with dual energy x-ray absorptiometry (DEXA), carotid intima media thickness (CIMT) measured by ultrasound, and hepatic triglyceride content measured using magnetic resonance (MR) imaging-estimated proton density fat fraction (PDFF). These measures allow for the early, noninvasive study of adiposity-related metabolic risk. The overall aim of this two-study research plan is to characterize the level of measurable risk using these sensitive markers in treated and untreated children with mental health disorders, and to evaluate the magnitude of change in risk that can be observed using these biomarkers in children receiving a well established behavioral weight-loss intervention.

DETAILED DESCRIPTION:
This project will utilize sensitive, early biomarkers of disease risk, including whole body adiposity with DEXA, PDDF and CIMT, directly relevant to diabetes and cardiovascular disease risk. The primary goals of this study are to deliver an evidence-based weight loss intervention to the population of youth who are overweight or obese as a result of antipsychotic treatment, to characterize metabolic risk associated with weight using sensitive biomarkers, and to evaluate the magnitude of change observed in these biomarkers in children receiving an established behavioral weight-loss intervention.

Aim 1: To evaluate the main effect of time of 16 weeks of a Behavioral Weight Loss (BWL) intervention on DEXA-measured whole body adiposity in overweight/obese antipsychotic (AP)-treated children compared to nonpsychiatric (NP) overweight or obese healthy controls, and in AP-treated youth randomized to monthly Usual Care (UC).

Aim 2: To evaluate the main effect of time of 16 weeks of a BWL intervention on PDFF in overweight/obese AP-treated children compared to NP overweight or obese healthy controls, and in AP-treated youth randomized monthly UC.

Aim 3: To evaluate the main effect of time of 16 weeks of a weekly behavioral weight loss intervention on CIMT in overweight/obese AP-treated children compared to NP overweight or obese healthy controls, and in AP-treated youth randomized monthly UC.

ELIGIBILITY:
INCLUSION CRITERIA

* 6-18 years old (at any point during study participation)
* BMI percentile > 85
* Meet DSM-IV criteria for one or more childhood onset psychiatric disorders including disruptive behavior disorders (attention deficit disorder, conduct disorder, oppositional defiant disorder and disruptive behavior disorder not otherwise specified), affective disorders (bipolar affective disorder, major depressive disorder and mood disorder not otherwise specified), anxiety disorders (generalized anxiety disorder, obsessive compulsive disorder, separation anxiety, social and other specific phobias) as well as other disorders, including autism spectrum disorders (autistic disorder, Asperger's Syndrome and pervasive developmental disorder not otherwise specified), psychotic disorders (schizophreniform disorder, schizophrenia and psychotic disorder not otherwise specified) and movement disorders (tic disorder, Tourette's Syndrome) as determined by semi-structured diagnostic interview (EXCEPT for the Obese or Overweight Control Group, none of whom can meet criteria for any DSM-IV Axis I psychiatric illness)
* Currently treated with an atypical antipsychotic medication (EXCEPT for the Obese or Overweight Healthy Control Group, none of whom can be treated with any psychotropic medications Participants treated with any psychotropic medication may not have any medication changes for 1 month prior to study enrollment at the discretion of the PI, and Antipsychotic-Treated Participants must be treated with an antipsychotic > approximately 12 weeks with no antipsychotic medication dose changes for 1 month
* The Healthy Overweight or Obese Control Group may not be currently taking any prescription medications (multivitamins, over the counter medications, glucocorticoid nasal spray and inhalers are permitted, as well as non-sedating antihistamines such as but not limited to Claritin (loratadine) and Zyrtec (cetirizine)
* Participants between 6-17 years old will be able to give assent and have a parent/guardian that can provide written informed consent, and 18 year-old participants will be able to provide written informed consent.

EXCLUSION CRITERIA

* Do not meet DSM-IV criteria for any Axis I psychiatric illness per PI discretion (EXCEPT for Overweight or Obese Healthy reference group)
* Any lifetime use of antipsychotics (EXCEPT for Antipsychotic-Treated Participants, with the individuals in the latter group possibly having a remote, brief prior antipsychotic exposure that may be considered for enrollment on a case by case basis by the PI)
* The presence of any serious medical disorder that may confound the assessment of relevant biologic measures or diagnoses, including: significant organ system dysfunction; endocrine disease, including type 1 or type 2 diabetes mellitus; coagulopathy; anemia; or acute infection; all based on PI discretion Participants regularly taking within the last 3 months any glucose lowering agent, lipid lowering agent, exogenous testosterone, recombinant human growth hormone, or any other endocrine agent that might confound substrate metabolism, oral glucocorticoids (glucocorticoid nasal spray and inhalers are permitted), sedating antihistamines (non-sedating antihistamines such as but not limited to Claritin (loratadine) and Zyrtec (cetirizine) are permitted), and certain mood stabilizing agents including antiepileptic medications (lamotrigine is permitted) and Lithium, as these medications may themselves worsen or otherwise alter weight gain, glucose and lipid regulation or otherwise make it difficult to assess the effects of the antipsychotic alone; (note that exposure to many psychotropic agents including stimulants, SSRI's and SNRI's are permitted in the Antipsychotic-Treated and Non-Antipsychotic Treated Groups in Study 1 in order to maintain the generalizability of the sample)
* IQ < 70 (based on school records and/or evaluation by clinician and at the discretion of the PI)
* Current DSM IV diagnosed substance abuse or dependence
* Past history of, or current dyskinesia
* Stimulant dosage significantly higher (per PI judgment) than the equivalent of approximately 2 mg/kg/day methylphenidate equivalent dose (EXCEPT in the Obese or Overweight Control Group, none of whom can be taking stimulant medications)
* Unable to provide assent or informed consent
* Active suicidality or a primary diagnosis of depression
* Unwilling to allow study staff to contact subject's primary care physician to alert to any significant, abnormal clinical findings or test results obtained as part of study participation

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ginger E Nicol, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nicol GE, Kolko R, Lenze EJ, Yingling MD, Miller JP, Ricchio AR, Schweiger JA, Findling RL, Wilfley D, Newcomer JW. Adiposity, Hepatic Triglyceride, and Carotid Intima Media Thickness During Behavioral Weight Loss Treatment in Antipsychotic-Treated Youth: A Randomized Pilot Study. J Child Adolesc Psychopharmacol. 2019 Aug;29(6):439-447. doi: 10.1089/cap.2018.0120. Epub 2019 Apr 17. PMID 30994376

RESULTS

PARTICIPANT FLOW:
Groups:
- Antipsychotic Treated Educational Control: Antipsychotic treated participants randomized to this arm will receive diet and exercise education at monthly intervals with a study clinician or coordinator.
  Diet and Exercise Education: Participants assigned to this arm will receive monthly medically validated, individualized diet and exercise education by a trained research professional.
- Antipsychotic Treated Weekly Behavioral Weight Loss: Antipsychotic treated participants randomized to this arm will engage in an evidence-based, 16 week manualized behavioral weight loss intervention that includes weekly meetings and phone check-ins with a trained study therapist.
  Behavioral Weight Loss: This intervention is a family-based, behavioral weight loss program that has been employed in studies with overweight and obese children, as well as with children who have diabetes. For the proposed study, the program has been modified to fit the needs of disruptive and behaviorally disturbed youth and their families. The modified program includes 16 weeks of weekly visits with a study interventionist, and supplemental phone contacts as needed. Phone contacts will only replace in-person visits if absolutely necessary to achieve the visit.
- Non-antipsychotic Treated Weekly Behavioral Weight Loss: Participants assigned to this arm will engage in an evidence-based, 16 week manualized behavioral weight loss intervention that includes weekly meetings and phone check-ins with a trained study therapist.
  Behavioral Weight Loss: This intervention is a family-based, behavioral weight loss program that has been employed in studies with overweight and obese children, as well as with children who have diabetes. For the proposed study, the program has been modified to fit the needs of disruptive and behaviorally disturbed youth and their families. The modified program includes 16 weeks of weekly visits with a study interventionist, and supplemental phone contacts as needed. Phone contacts will only replace in-person visits if absolutely necessary to achieve the visit.
Period: Overall Study
Arm/Group | Antipsychotic Treated Educational Control | Antipsychotic Treated Weekly Behavioral Weight Loss | Non-antipsychotic Treated Weekly Behavioral Weight Loss
Started | 7 | 19 | 21
Completed | 6 | 15 | 17
Not Completed | 1 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Antipsychotic Treated Educational Control | Antipsychotic Treated Weekly Behavioral Weight Loss | Non-antipsychotic Treated Weekly Behavioral Weight Loss | Total
Number analyzed (Participants) | 7 | 19 | 21 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.80 (2.21) | 13.35 (2.57) | 13.42 (2.46) | 13.30 (2.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 15 | 21
  Male | 6 | 14 | 6 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 7 | 19 | 20 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 6 | 9
  White | 7 | 15 | 13 | 35
  More than one race | 0 | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Primary Diagnosis [Count of Participants; unit: Participants]
  Autism | 4 | 11 | 0 | 15
  Pervasive Development Disorder (PDD) | 1 | 0 | 0 | 1
  Attention Deficit Hyperactivity Disorder (ADHD) | 1 | 4 | 0 | 5
  Mood Disorder | 1 | 2 | 0 | 3
  Anxiety Disorder | 0 | 1 | 0 | 1
  Psychosis | 0 | 1 | 0 | 1
Height [Mean (Standard Deviation); unit: meters] | 1.58 (0.17) | 1.58 (0.15) | 1.63 (0.11) | 1.60 (0.14)
Weight [Mean (Standard Deviation); unit: kilograms] | 72.37 (16.11) | 77.08 (32.60) | 85.76 (23.07) | 80.26 (26.62)
DEXA-Measured Body Composition [Mean (Standard Deviation); unit: percentage of body composition]
  DEXA Total Percent Fat | 45.40 (6.76) | 41.76 (8.53) | 42.24 (5.38) | 42.51 (6.97)
  DEXA Total Percent Lean | 52.12 (6.81) | 55.48 (8.23) | 55.01 (5.15) | 54.77 (6.73)
Proton Density Fat Fraction (PDFF) [Mean (Standard Deviation); unit: percentile] | 12.01 (7.82) | 6.52 (8.21) | 4.72 (8.61) | 6.58 (8.54)
Carotid Intima Media Thickness [Mean (Standard Deviation); unit: centimeters] | 0.0494 (0.0058) | 0.0451 (0.0074) | 0.0504 (0.0065) | 0.0484 (0.0070)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter-squared] | 28.72 (2.09) | 29.70 (6.83) | 31.86 (5.25) | 30.52 (5.69)
Body Mass Index (BMI) Percentile [Mean (Standard Deviation); unit: percentile] | 97.77 (1.03) | 96.55 (3.30) | 97.69 (2.16) | 97.24 (2.60)
Body Mass Index (BMI) Z-Score [Mean (Standard Deviation); unit: z-score] — The BMI Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population (i.e., healthy, age and sex-matched children). Negative numbers indicate values lower than the reference population and positive numbers indicate values higher than the reference population.
  z-score | 2.05 (0.23) | 1.99 (0.47) | 2.13 (0.38) | 2.06 (0.40)
Waist Circumference [Mean (Standard Deviation); unit: centimeters] | 99.86 (10.35) | 99.45 (19.35) | 102.40 (16.07) | 100.83 (16.58)
Baseline Fasting Laboratory Values [Mean (Standard Deviation); unit: mg/dl]
  Glucose | 93.71 (10.01) | 91.32 (7.42) | 87.62 (4.99) | 90.02 (7.13)
  Total Cholesterol | 170.14 (9.67) | 169.47 (37.55) | 157.81 (29.09) | 164.36 (31.10)
  Triglycerides | 114.43 (44.49) | 106.26 (59.11) | 99.14 (61.30) | 104.30 (57.35)
  HDL Cholesterol | 45.00 (6.16) | 46.95 (10.20) | 50.71 (10.74) | 48.34 (10.04)
  LDL Cholesterol | 102.29 (10.95) | 101.68 (27.32) | 87.24 (23.40) | 95.32 (24.49)
Aberrant Behavior Checklist (ABC) [Mean (Standard Deviation); unit: units on a scale] — This instrument is a five-factor scale comprising 58 items under the categories of (I) Irritability, Agitation, Crying; (II) Lethargy, Social Withdrawal; (III) Stereotypic Behavior; (IV) Hyperactivity, Noncompliance; and (V) Inappropriate Speech. The 15-item Irritability subscale score ranges from 0 to 45. The cut-off of ≥ 18 on this subscale will identify individuals that are 1.3 to 1.5 SD above the mean. A lower score is better.The total score can range from a minimum of 0 (no problem behaviors) to a maximum of 174, with higher scores indicating a worse outcome/more symptoms.
  units on a scale
    Total Score | 53.43 (20.14) | 35.61 (24.29) | 6.81 (13.39) | 25.17 (26.11)
    Irritability | 18.57 (8.75) | 11.06 (8.30) | 2.19 (4.81) | 8.15 (9.13)
Child Behavior Checklist (CBCL) [Mean (Standard Deviation); unit: units on a scale] — The CBCL/ABCL is a 113 item scale that serves as a general screening measure of behavior problems, competencies, and school functioning. Each item is scored a 0, 1, or 2. A lower score is better. The eight empirically-based syndrome scales are: Aggressive Behavior, Anxious/Depressed, Attention Problems, Rule-Breaking Behavior, Somatic Complaints, Social Problems, Thought Problems and Withdrawn/Depressed.
  units on a scale | 70.14 (26.34) | 57.06 (28.39) | 16.67 (15.20) | 40.61 (31.80)

OUTCOME MEASURES:

1. Primary Outcome: DEXA-measured Adiposity
Description: Dual-Energy X-Ray Absorptiometry (DEXA) will be used to assess body fat at baseline and following 16 weeks of participation in a behavioral weight loss intervention.
Time Frame: Baseline and 16 weeks
Population: Modified Intent to Treat (ITT) sample with week 0 and week 16 data.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Antipsychotic Treated Educational Control | Antipsychotic Treated Weekly Behavioral Weight Loss | Non-antipsychotic Treated Weekly Behavioral Weight Loss
Number analyzed (Participants) | 6 | 15 | 17
kilograms | 0.76 (2.05) | -0.43 (3.13) | -2.79 (3.35)
Statistical Analysis 1: Comparison: Antipsychotic Treated Educational Control vs Antipsychotic Treated Weekly Behavioral Weight Loss vs Non-antipsychotic Treated Weekly Behavioral Weight Loss; An ANCOVA was used to test for differences between groups at endpoint, controlling for baseline values; Test type: Superiority; p = 0.01, ANCOVA — The p-value refers to the treatment group term in the model. The a priori threshold for statistical significance in this planned primary test was p < 0.05

2. Primary Outcome: Proton Density Fat Fraction (PDFF)
Description: 1H Magnetic Resonance Spectroscopy (MRS) of liver will be used to assess intracellular triglyceride content at baseline and following 16 weeks of participation in a behavioral weight loss intervention.
Time Frame: Baseline and 16 weeks
Population: Modified Intent to Treat (ITT) sample with week 0 and week 16 data.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Antipsychotic Treated Educational Control | Antipsychotic Treated Weekly Behavioral Weight Loss | Non-antipsychotic Treated Weekly Behavioral Weight Loss
Number analyzed (Participants) | 6 | 12 | 16
percent | -0.62 (1.57) | -0.41 (4.95) | -1.75 (4.93)
Statistical Analysis 1: Comparison: Antipsychotic Treated Educational Control vs Antipsychotic Treated Weekly Behavioral Weight Loss vs Non-antipsychotic Treated Weekly Behavioral Weight Loss; An ANCOVA was used to test for differences between groups at endpoint, controlling for baseline values; Test type: Superiority; p = 0.04, ANCOVA — [p-value comment as in outcome 1, analysis 1]

3. Primary Outcome: Carotid Artery Intima Media Thickness (CIMT)
Description: 9-13-MHZ B-mode Carotid Ultrasound will be used to assess intima media thickness at baseline and following 16 weeks of participation in a behavioral weight loss intervention.
Time Frame: Baseline and 16 weeks
Population: Modified Intent to Treat (ITT) sample with week 0 and week 16 data.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Antipsychotic Treated Educational Control | Antipsychotic Treated Weekly Behavioral Weight Loss | Non-antipsychotic Treated Weekly Behavioral Weight Loss
Number analyzed (Participants) | 6 | 10 | 17
millimeters | -0.0014 (0.0045) | 0.0032 (0.0098) | 0.0004 (0.0064)
Statistical Analysis 1: Comparison: Antipsychotic Treated Educational Control vs Antipsychotic Treated Weekly Behavioral Weight Loss vs Non-antipsychotic Treated Weekly Behavioral Weight Loss; An ANCOVA was used to test for differences between groups at endpoint, controlling for baseline values; Test type: Superiority; p = 0.70, ANCOVA — [p-value comment as in outcome 1, analysis 1]

4. Other Pre Specified Outcome: Aberrant Behavior Checklist (ABC)
Description: Change From Baseline in Aberrant Behavior Checklist - Irritability Subscale at 16 Weeks
Time Frame: Baseline and 16 weeks
Population: Modified Intent to Treat (ITT) sample with week 0 and week 16 data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Antipsychotic Treated Educational Control | Antipsychotic Treated Weekly Behavioral Weight Loss | Non-antipsychotic Treated Weekly Behavioral Weight Loss
Number analyzed (Participants) | 6 | 15 | 16
units on a scale | 3.00 (4.65) | -1.27 (5.82) | -1.38 (4.32)
Statistical Analysis 1: Comparison: Antipsychotic Treated Educational Control vs Antipsychotic Treated Weekly Behavioral Weight Loss vs Non-antipsychotic Treated Weekly Behavioral Weight Loss; An ANCOVA was used to test for differences between groups at endpoint, controlling for baseline values; Test type: Superiority; p = 0.003, ANCOVA — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a period of 16 weeks.
Arm/Group | Antipsychotic Treated Educational Control | Antipsychotic Treated Weekly Behavioral Weight Loss | Non-antipsychotic Treated Weekly Behavioral Weight Loss
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 0/7 | 0/19 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-04): https://cdn.clinicaltrials.gov/large-docs/94/NCT01222494/Prot_SAP_000.pdf